CLINICAL TRIAL: NCT02580487
Title: Perioperative Pain Management of Pediatric Appendectomy Patients in Kuopio University Hospital During the Years 2010-2012
Brief Title: Perioperative Pain Management of Pediatric Appendectomy Patients
Acronym: umpikipu
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Other Study IDs: KUH01012012
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Appendicitis
Keywords: acute appendicitis; pain management; analgesics; pediatric patients; laparoscopy; open surgery
MeSH Terms: conditions — Appendicitis; Agnosia | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- retrospective group: Patients whose pain evaluation, analgesics used and details of surgery were collected from patient files
  Interventions: Procedure: appendicectomy
- Prospective group: Patients who were interviewed before and after surgery when they were at the hospital
  Interventions: Procedure: appendicectomy

INTERVENTIONS:
Procedure: appendicectomy — Appendix was removed either laparoscopically or open surgery

SUMMARY:
Acute appendicitis is the most common illness that brings pediatric patients to the hospital for surgical treatment. Abdominal pain is the symptom because of which the patients go to the hospital. Some patients have severe pain and need analgesics before the final diagnosis and before surgery. After surgery most patient experience pain and at least 80 % of the patients need postoperative pain medication. For two decades there has been a clinical guideline for pain management in Kuopio University Hospital (KUH). The investigators aim was to evaluate how well the pain management for pediatric patient works in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* In prospective patients informed consent obtained
* Appendectomy performed

Exclusion Criteria:

* No informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 152 pediatric patients that were operated on in KUH during the years 2010-2012 due to acute appendicitis.
  In addition we assessed 26 pediatric appendectomy patients and their pain at rest, when coughing and when compressing the wound area propsectively when they were at hospital
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pain | from preoperative evaluation until the patient left hospital maximum of 7 days
  pain is asked preoperatively and at the first postoperative day measured with numeral rating scale

SECONDARY OUTCOMES:
amount of opioids used during hospital stay | from preoperative evaluation until the patient left hospital maximum of 7 days
  collected from patient files

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland